CLINICAL TRIAL: NCT00920517
Title: Safety and Immunogenicity of a 2-Dose Regimen of rDEN2/4Δ30 Dengue Vaccine With Boosting at 4 Versus 6 Months
Brief Title: Safety and Immune Response to Two Doses of rDEN2/4delta30 Dengue Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIR 250
Record Dates: First submitted 2009-06-11; First posted 2009-06-15 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants will receive 1 injection of rDEN2/4delta30(ME) or placebo vaccine on Days 0 and 180
  Interventions: Biological: rDEN2/4delta30(ME) vaccine; Biological: Placebo
- 2 (Active Comparator): Participants will receive 1 injection of rDEN2/4delta30(ME) or placebo vaccine on Days 0 and 120
  Interventions: Biological: rDEN2/4delta30(ME) vaccine; Biological: Placebo

INTERVENTIONS:
Biological: rDEN2/4delta30(ME) vaccine — 10^3 PFU dose
Biological: Placebo — placebo for rDEN2/4delta30(ME) vaccine

SUMMARY:
Dengue fever, caused by dengue viruses, is a major health problem in the tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses, which cause dengue fever and dengue shock syndrome, are a major cause of morbidity and mortality in several of the world's tropical and subtropical regions. The rDEN2/4delta30(ME) vaccine is a live attenuated dengue virus vaccine that may be protective against dengue virus serotype 2 (DEN2). The purpose of this study is to evaluate the safety and immunogenicity of the rDEN2/4delta30(ME) vaccine in healthy adults.

This study will last approximately 5 to 7 months with 25 study visits. Participants will be randomly assigned into one of two cohorts. Participants in Cohort 1 will receive an injection of rDEN2/4delta30(ME) or placebo vaccine at Days 0 and 180. Participants in Cohort 2 will receive an injection of rDEN2/4delta30(ME) or placebo vaccine at Days 0 and 120. Participants will be asked to record their temperature in a diary for 16 days after each vaccination. At each study visit a physical examination, symptom history, and blood and urine collection will occur.

ELIGIBILITY:
Inclusion Criteria:

* Good general health as determined by means of the screening procedures.
* Available for the duration of the study (32 weeks for cohort 1 and 23 weeks for cohort 2)
* Willing to use effective methods of contraception

Exclusion Criteria:

* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator will affect the ability of the volunteer to understand and cooperate with the requirements of the study protocol
* Neutropenia as defined by an ANC ≤1500/mm3
* ALT level above the laboratory-defined upper limit of normal
* Serum creatinine level above the laboratory-defined upper limit of normal
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* Positive HIV-1 serology by screening and confirmatory assays
* Positive for hepatitis C virus (HCV) by screening and confirmatory assays
* Positive hepatitis B surface antigen (HBsAg) by enzyme-linked immunosorbent assay (ELISA)
* Known immunodeficiency syndrome
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study
* Receipt of a live vaccine within the 4 weeks or a killed vaccine within the 2 weeks prior to entry into the study
* Has had spleen surgically removed
* Receipt of blood products within the 6 months prior to study entry
* History or serologic evidence of previous dengue virus infection or other flavivirus infection (e.g. yellow fever virus, St. Louis encephalitis, West Nile virus).
* Previous receipt of yellow fever or dengue vaccine (licensed or experimental)
* Persons who have received any investigational agent in the 30 days prior to study entry
* Persons who have definite plans to travel to a dengue endemic area during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Determine the frequency of vaccine related AEs for each dose, graded by severity. | Throughout study
Compare the immunogenicity of the two 2-dose regimens of the rDEN2/4Δ30(ME) candidate vaccine as assessed by neutralizing antibody titers to DEN2 | At 4 and 6 weeks after each vaccination

SECONDARY OUTCOMES:
Assess the frequency, quantity, and duration of viremia after each dose of vaccine. | Throughout study
Determine the number of vaccinees infected with rDEN2/4Δ30(ME) | Throughout study
Comparison of infectivity rates, safety, and immunogenicity between dose 1 and dose 2 withhin cohort and between cohorts | Throughout study
Evaluation of the phenotype and activation of peripheral blood mononuclear cells at primary infection and upon reinfection with the DEN2/4Δ30(ME) vaccine. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Center for Immunization Research, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Katzelnick LC, Fonville JM, Gromowski GD, Bustos Arriaga J, Green A, James SL, Lau L, Montoya M, Wang C, VanBlargan LA, Russell CA, Thu HM, Pierson TC, Buchy P, Aaskov JG, Munoz-Jordan JL, Vasilakis N, Gibbons RV, Tesh RB, Osterhaus AD, Fouchier RA, Durbin A, Simmons CP, Holmes EC, Harris E, Whitehead SS, Smith DJ. Dengue viruses cluster antigenically but not as discrete serotypes. Science. 2015 Sep 18;349(6254):1338-43. doi: 10.1126/science.aac5017. PMID 26383952